CLINICAL TRIAL: NCT06614244
Title: Randomized Multicenter Trial of Oral Immunotherapy for Food Protein Induced Enterocolitis Syndrome
Brief Title: Oral Immunotherapy for Food Protein Induced Enterocolitis Syndrome
Acronym: DOPAxSEA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6563
Record Dates: First submitted 2024-09-02; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: FPIES
MeSH Terms: interventions — Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DOPA group (Experimental): Children affected by acute persistent FPIES subjected to OIT for the offending food
  Interventions: Procedure: Oral immunotherapy (OIT)
- Diet group (Active Comparator): Children affected by acute persistent FPIES subjected to the traditional measure, i.e. the elimination diet for the offending food
  Interventions: Dietary Supplement: Culprit food elimination diet

INTERVENTIONS:
Procedure: Oral immunotherapy (OIT) — OIT in DOPA group will be implemented as follows. Both the first micro-dose of the offending food and the subsequent micro-increments will be administered at home. Any interruptions and resumptions of OIT, due to intercurrent events (e.g. infections), will be managed via email with or without medical visit via video call. Patients will be provided with ondansetron (sublingual film) and instructions for its use. An explanatory letter will also be provided in case of need for emergency room access.
  Arms: DOPA group
Dietary Supplement: Culprit food elimination diet — The Diet group consists of a population of children affected by acute persistent FPIES subjected to the traditional measure, i.e. the elimination diet of the incriminated food.
  Arms: Diet group

SUMMARY:
Food Protein Induced Enterocolitis Syndrome (FPIES) is a food allergy characterized by clinical manifestations of varying severity that can be, very rarely, severe to the point of leading to shock. Acute FPIES is nowaday the most common presentation of the disease. It is characterized by repeated, projectile vomiting (usually arising between 1 and 4 hours after ingestion of the culprit food) accompanied by pallor, hypotonia, and lethargy, with complete resolution of the aforementioned symptoms almost always within a few hours. Dietary management of FPIES currently involves avoiding allergens, offering complementary foods to encourage normal growth and providing families with individualized feeding plans. The elimination diet does not promote healing, it only prevents adverse reactions from culprit food ingestion. Recovery (i.e. tolerance to the culprit food) is achieved spontaneously over time. However, for some children, tolerance does not occur. These patients suffer from persistent FPIES. For these patients oral immunotherapy (OIT) is not yet planned and randomized and controlled studies are needed to demonstrate its efficacy and safety. The primary objective of the study will be to verify, with a multicenter, prospective, randomized study, stratified for the main 4 offending foods in Italy (cows milk, hens egg, fish and cereals), open-label and with an adequate sample size, the efficacy and safety of an OIT procedure in children affected by acute persistent FPIES. The comparison will be made between a population of children affected by acute persistent FPIES subjected to OIT for the offending food (DOPA group) and a population of children affected by acute persistent FPIES subjected to the traditional measure, i.e. the elimination diet for the offending food (Diet group).

Efficacy will be measured through:

* Comparison of the percentages of children who have increased their reactivity threshold even to the point of no adverse reactions to the offending food following the intake of a normal dose for their age in the two populations during treatment;
* Comparison of the percentages of children who have reached tolerance towards the culprit food in the two populations;

Safety will be measured through:

- Comparison of the percentages of children who have presented adverse reactions following the ingestion (accidental in the Diet group and expected in the DOPA group) of the culprit food after enrollment in the study.

The definitions of desensitization and tolerance are taken from the EAACI 2018 guidelines on immunotherapy for IgE-mediated AA. In particular, desensitization corresponds to the absence of adverse reactions following the ingestion of the culprit food (in quantities up to a normal dose for age) during oral immunotherapy. This is a reversible or partially reversible clinical response that depends on continued exposure to the allergen. If the administration of the allergen is interrupted, the previous level of clinical reactivity may return. Tolerance corresponds to the absence of adverse reactions following the ingestion of the culprit food despite a period of absence of exposure.

ELIGIBILITY:
Inclusion criteria

* Pediatric patients (under 18 years of age) affected by persistent acute food protein-induced enterocolitis syndrome.
* The last anamnestic acute episode must not be more than 1 month prior to the date of inclusion in the study. The anamnestic definition of acute episode will be based on the use of Miceli Sopo 2022 questionnaire for food protein-induced enterocolitis syndrome. In case it is not clear whether the disease is active or not, an oral food challenge will be performed to verify the possible acquisition of tolerance (a procedure that is part of the routine management for this allergy). Inclusion in the study must occur within 1 month of the possible failure of the aforementioned oral food challenge. Regarding patients with multiple FPIES (expected to be approximately 6% of the total patients included, a small minority), OIT will be started for the nutritionally most relevant food among those eligible.

Exclusion criteria

* Absence of inclusion criteria.
* Transition from acute FPIES to IgE-mediated AA.
* Absence of informed consent approval by their caregivers.
* Failure to use email by their caregivers.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the percentages of participants who will achieve desensitization to the culprit food in the two populations | 18 months
  Efficacy will be measured through comparison of the percentages of children who will have increased their threshold of reactivity to the incriminated food following the intake of a normal dose for their age, in the two study populations (Definition of desensitization and tolerance according to EAACI 2018 guidelines on immunotherapy for IgE-mediated AA)

SECONDARY OUTCOMES:
Phenotypic characteristics of the patient who responds to OIT | 18 months
  Define the phenotypic characteristics of the patient with acute FPIES who will respond best to OIT

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Miceli Sopo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Pediatria, Roma, Italy